CLINICAL TRIAL: NCT07198672
Title: A Multicenter, Single-arm, Exploratory Clinical Study of Herombopag Olamine Tablets for the Primary Prevention of Treatment-related Thrombocytopenia in HER2-positive Breast Cancer Patients Receiving T-DM1 Therapy
Brief Title: Primary Prevention of Thrombocytopenia Associated With T-DM1 Therapy in HER2 Positive Breast Cancer With Herombopag
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhenzhen Liu (Other Government)
Responsible Party: Sponsor-Investigator, Zhenzhen Liu, Clinical Professor, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HN-CTIT-HQ-001
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Herombopag Group (Experimental): Preventive treatment with eltrombopag should be initiated on the evening of the first day of each T-DM1 treatment cycle (typically 3 weeks). Eltrombopag 7.5 mg (initial dose) should be administered orally once daily for a maximum duration of 21 days.
  Interventions: Drug: Herombopag

INTERVENTIONS:
Drug: Herombopag — Each T-DM1 treatment cycle typically lasts 3 weeks, with prophylactic administration of eltrombopag continuing until 21 days after the end of that T-DM1 treatment cycle. Oral administration of eltrombopag ethanolamine tablets begins on the evening of the first day of each T-DM1 treatment cycle, starting at a dose of 7.5 mg once daily.

SUMMARY:
Ado-trastuzumab emtansine (T-DM1) demonstrates favorable efficacy in breast cancer treatment but is frequently associated with thrombocytopenia. Multiple studies indicate that Asian populations face a higher risk of developing thrombocytopenia during T-DM1 therapy, with incidence rates ranging from 52.5% to 69.8% and ≥Grade 3 rates between 29.8% and 45.0%. Severe thrombocytopenia not only increases bleeding risks but may also necessitate T-DM1 dose delays or reductions, thereby compromising treatment efficacy and diminishing patient survival and quality of life. Herombopag selectively binds to the transmembrane region of TPO-R, activating TPO-R-dependent STAT and MAPK signaling pathways. This effectively stimulates megakaryocyte proliferation and differentiation, promoting thrombopoiesis. However, high-level evidence supporting the use of Herombopag for primary prevention of T-DM1-induced thrombocytopenia in breast cancer remains lacking.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥18 years;
2. Histopathologically or cytologically confirmed diagnosis of breast cancer;
3. Tumor tissue confirmed as HER2-positive, defined as immunohistochemistry (IHC) showing +++, or IHC++ with fluorescence in situ hybridization (FISH) demonstrating HER2-positive status;
4. Planned to receive T-DM1 regimen based on clinical judgment;
5. ECOG PS score: 0-2;
6. Expected survival greater than 12 weeks;
7. Adequate organ and bone marrow function.

Exclusion Criteria:

1. A confirmed history of severe allergic reactions to the active ingredients or excipients of the therapeutic drug;
2. Presence of other underlying diseases or comorbidities causing thrombocytopenia, such as aplastic anemia, immune thrombocytopenia, myelodysplastic syndrome, etc.;
3. Individuals with hereditary bleeding disorders, coagulation dysfunction, high bleeding risk, or a history of thrombotic events (e.g., transient ischemic attack, cerebral hemorrhage, cerebral infarction, pulmonary embolism) within 6 months prior to initial medication use;
4. Individuals with uncontrolled hypertension and a history of hypertensive crisis or hypertensive encephalopathy;
5. Pregnant or lactating women;
6. Presence of multiple factors affecting oral drug absorption, such as dysphagia, nausea/vomiting, chronic diarrhea, or intestinal obstruction;
7. History of severe psychiatric disorders, substance abuse, alcoholism, or drug addiction;
8. Currently participating in interventional clinical research treatment, or having received other investigational drugs or devices within 4 weeks prior to first dosing (individuals who failed screening for other clinical trials may be included in this study);
9. Any other factors deemed by the investigator to increase study risk, affect patient compliance with the protocol, or impact the patient's ability to complete the trial, such as physiological or psychological conditions that make participation in this study inappropriate;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of thrombocytopenia (<100 × 10⁹/L) | up to 6 cycles (each cycle is 21 days)
  PLT <100 × 10⁹/L

SECONDARY OUTCOMES:
The time of the first occurrence of thrombocytopenia (<100 × 10⁹/L); | up to 6 cycles (each cycle is 21 days)
  Time at which PLT < 100 × 10⁹/L occurs
Incidence of AEs | up to 6 cycles (each cycle is 21 days)
  Record the occurrence of adverse events during the study period

IPD SHARING:
Plan to Share IPD: No